CLINICAL TRIAL: NCT06344832
Title: Somatostatin Receptor Antagonist PET/CT for Pre-operative N Stage Evaluation in Patients With Gastro-entero-pancreatic Neuroendocrine Tumors
Brief Title: SSTR PET/CT for Preoperative N Stage Evaluation in GEP-NETs
Status: Not yet recruiting | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: K5098
Record Dates: First submitted 2024-03-28; First posted 2024-04-03 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-03

CONDITIONS: Gastro-entero-pancreatic Neuroendocrine Tumor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The research aims to prospectively include patients with GEP-NENs, undergo preoperative imaging assessment (including PET/CT and contrast-enhanced CT), and accurately delineate lymph node regions. Through postoperative pathological reports, the diagnostic performance of lymph node metastasis (LNM) in GEP-NENs is evaluated. Factors influencing the diagnostic accuracy of SSTR-PET/CT and contrast-enhanced CT are also investigated.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years old;
2. Patients diagnosed with GEP-NEN by surgical pathology;
3. Complete medical records including basic information and treatment process;
4. Patients who have undergone preoperative contrast-enhanced CT and 68Ga-SSTR-PET/CT, and have consented to the 68Ga-SSTR-PET/CT project in the Nuclear Medicine Department.

Exclusion Criteria:

1. Presence of concomitant malignancies;
2. Cases diagnosed pathologically as non-GEP-NEN.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with GEP-NEN undergoing surgical treatment at Peking Union Medical College Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2028-03-01 (Estimated); Study Completion 2030-03-01 (Estimated)

PRIMARY OUTCOMES:
lymph node metastasis status | 2024.04.01~2030.03.01
  lymph node metastasis status confirmed by histopathology